CLINICAL TRIAL: NCT03015532
Title: A Phase 2b, Randomized, Double-Blind, Saline Placebo- and Active-Controlled, Multicenter Study of HTX-011 Via Infiltration for Postoperative Analgesia in Subjects Undergoing Total Knee Arthroplasty
Brief Title: Total Knee Arthroplasty Infiltration Study for Postoperative Analgesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTX-011-209
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Results first posted 2021-10-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain
Keywords: knee; knee replacement; arthroplasty; joint replacement; knee pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (8):
- Cohort 1, Group 1: HTX-011 (Experimental): HTX-011 (bupivacaine/meloxicam), 200 mg/6 mg via instillation
  Interventions: Drug: HTX-011
- Cohort 1, Group 2: HTX-011 (Experimental): HTX-011 (bupivacaine/meloxicam), 200 mg/6 mg via injection and instillation (combination)
  Interventions: Drug: HTX-011
- Cohort 1, Group 3: Saline Placebo (Placebo Comparator): Saline placebo via injection
  Interventions: Drug: Saline Placebo
- Cohort 1, Group 4: Bupivacaine HCI (Active Comparator): Bupivacaine HCl without epinephrine, 125 mg via injection
  Interventions: Drug: Bupivicaine HCl
- Cohort 2, Group 1: HTX-011 (Experimental): HTX-011 (bupivacaine/meloxicam), 400 mg/12 mg via instillation
  Interventions: Drug: HTX-011
- Cohort 2, Group 2: HTX-011 + Ropivacaine (Experimental): HTX-011 (bupivacaine/meloxicam), 400 mg/12 mg via instillation; Ropivacaine, 50 mg via injection
  Interventions: Drug: HTX-011; Drug: Ropivacaine
- Cohort 2, Group 3: Saline Placebo (Placebo Comparator): Saline placebo via injection
  Interventions: Drug: Saline Placebo
- Cohort 2, Group 4: Bupivacaine HCI (Active Comparator): Bupivacaine HCl without epinephrine, 125 mg via injection
  Interventions: Drug: Bupivicaine HCl

INTERVENTIONS:
Drug: HTX-011 — HTX-011 (bupivacaine/meloxicam), via instillation
  Arms: Cohort 1, Group 1: HTX-011; Cohort 1, Group 2: HTX-011; Cohort 2, Group 1: HTX-011; Cohort 2, Group 2: HTX-011 + Ropivacaine
Drug: Saline Placebo — Saline placebo via injection
  Arms: Cohort 1, Group 3: Saline Placebo; Cohort 2, Group 3: Saline Placebo
Drug: Bupivicaine HCl — Bupivacaine HCl without epinephrine
  Arms: Cohort 1, Group 4: Bupivacaine HCI; Cohort 2, Group 4: Bupivacaine HCI
Drug: Ropivacaine — Ropivacaine, via injection
  Arms: Cohort 2, Group 2: HTX-011 + Ropivacaine

SUMMARY:
This is a Phase 2b, randomized, double-blind, saline placebo- and active-controlled, multicenter study in subjects undergoing primary unilateral total knee arthroplasty (TKA) to evaluate the analgesic efficacy, safety, and pharmacokinetics (PK) of HTX-011 administered via infiltration to the surgical site.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled to undergo primary unilateral TKA under general anesthesia.
* Has not previously undergone TKA in either knee.
* Has an American Society of Anesthesiologists Physical Status of I, II, or III.
* Is able to demonstrate motor function by performing a timed 20-meter walk unassisted, but with the optional use of a 4-legged walker for balance.
* Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, sterile; or using acceptable contraceptives.

Exclusion Criteria:

* Has a planned concurrent surgical procedure (eg, bilateral TKA).
* Has a pre-existing concurrent acute or chronic painful/restrictive physical condition that may require analgesic treatment in the postoperative period for pain.
* Has a contraindication or a known or suspected history of hypersensitivity or idiosyncratic reaction to required study medications.
* Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months.
* Has taken NSAIDs within 10 days prior to the scheduled surgery.
* Has taken opioids within 24 hours prior to the scheduled surgery (3 days for long-acting).
* Has been administered bupivacaine within 5 days prior to the scheduled surgery.
* Has initiated treatment with medications within 1 month prior to study drug administration that can impact pain control.
* Has been administered systemic steroids within 5 half-lives or 10 days prior to administration of study drug.
* Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments.
* Has a known history of Hepatitis B, human immunodeficiency virus (HIV), or active Hepatitis C.
* Has uncontrolled anxiety, psychiatric, or neurological disorder that might interfere with study assessments.
* Has any chronic neuromuscular deficit of either femoral nerve function or thigh musculature. Has any chronic condition or disease that would compromise neurological or vascular assessments.
* Had a malignancy in the last year, with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half lives.
* Has undergone 3 or more surgeries within 12 months.
* Has a body mass index (BMI) >38 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Mobile, Alabama
  - Sheffield, Alabama
  - Phoenix, Arizona
  - La Jolla, California
  - Riverside, California
  - San Diego, California
  - Miami, Florida
  - Tamarac, Florida
  - Las Vegas, Nevada
  - Columbus, Ohio
  - Dayton, Ohio
  - Bellaire, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Webster, Texas

REFERENCES:
- [Derived] Lachiewicz PF, Lee GC, Pollak RA, Leiman DG, Hu J, Sah AP. HTX-011 Reduced Pain and Opioid Use After Primary Total Knee Arthroplasty: Results of a Randomized Phase 2b Trial. J Arthroplasty. 2020 Oct;35(10):2843-2851. doi: 10.1016/j.arth.2020.05.044. Epub 2020 May 27. PMID 32561266

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2, Group 1: HTX-011: HTX-011(bupivacaine/meloxicam), 400 mg/12 mg via instillation.
- Cohort 2, Group 2: HTX-011 + Ropivacaine: HTX-011(bupivacaine/meloxicam), 400 mg/12 mg via instillation; Ropivacaine, 50 mg via injection.
Period: Overall Study
Arm/Group | Cohort 1, Group 1: HTX-011 | Cohort 1, Group 2: HTX-011 | Cohort 1, Group 3: Saline Placebo | Cohort 1, Group 4: Bupivacaine HCI | Cohort 2, Group 1: HTX-011 | Cohort 2, Group 2: HTX-011 + Ropivacaine | Cohort 2, Group 3: Saline Placebo | Cohort 2, Group 4: Bupivacaine HCI
Started | 20 | 22 | 11 | 10 | 58 | 56 | 53 | 55
Completed | 20 | 22 | 11 | 10 | 58 | 54 | 51 | 55
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Group 1: HTX-011 | Cohort 1, Group 2: HTX-011 | Cohort 1, Group 3: Saline Placebo | Cohort 1, Group 4: Bupivacaine HCI | Cohort 2, Group 1: HTX-011 | Cohort 2, Group 2: HTX-011 + Ropivacaine | Cohort 2, Group 3: Saline Placebo | Cohort 2, Group 4: Bupivacaine HCI | Total
Number analyzed (Participants) | 20 | 22 | 11 | 10 | 58 | 56 | 53 | 55 | 285
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 17 | 5 | 4 | 31 | 34 | 36 | 38 | 177
  >=65 years | 8 | 5 | 6 | 6 | 27 | 22 | 17 | 17 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (7.52) | 58.6 (7.44) | 64.9 (4.64) | 65.3 (11.62) | 62.5 (8.63) | 63.2 (9.36) | 61.5 (8.31) | 61.4 (9.37) | 62.1 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 7 | 5 | 26 | 27 | 25 | 35 | 147
  Male | 7 | 13 | 4 | 5 | 32 | 29 | 28 | 20 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 3 | 1 | 9 | 16 | 12 | 16 | 74
  Not Hispanic or Latino | 13 | 12 | 8 | 9 | 49 | 40 | 41 | 39 | 211
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 2 | 3 | 6 | 5 | 8 | 7 | 39
  White | 15 | 18 | 9 | 7 | 51 | 49 | 45 | 47 | 241
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 11 | 10 | 58 | 56 | 53 | 55 | 285

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) Pain Intensity Scores at Rest (NRS-R) Through 48 Hours Postsurgery (AUC0-48).
Description: Pain intensity is assessed at rest using an 11-point NRS (0-10) where 0 represents "no pain" and 10 represents "worst pain imaginable" (using windowed worst observation carried forward to adjust for opioid rescue medication use). The theoretical range of AUC0-48 is 0-480.
Time Frame: 48 hours
Population: ITT Population
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Cohort 1, Group 1: HTX-011 | Cohort 1, Group 2: HTX-011 | Cohort 1, Group 3: Saline Placebo | Cohort 1, Group 4: Bupivacaine HCI | Cohort 2, Group 1: HTX-011 | Cohort 2, Group 2: HTX-011 + Ropivacaine | Cohort 2, Group 3: Saline Placebo | Cohort 2, Group 4: Bupivacaine HCI
Number analyzed (Participants) | 20 | 22 | 11 | 10 | 58 | 56 | 53 | 55
pain intensity score*hr | 386.12 (82.930) | 391.56 (84.450) | 405.82 (97.549) | 347.56 (103.422) | 322.08 (99.669) | 307.25 (127.674) | 396.36 (77.468) | 352.74 (100.887)

2. Secondary Outcome: Mean Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) Pain Intensity Scores at Rest (NRS-R) Through 72 Hours Postsurgery (AUC0-72).
Description: Pain intensity is assessed at rest using an 11-point NRS (0-10) where 0 represents "no pain" and 10 represents "worst pain imaginable" (using windowed worst observation carried forward to adjust for opioid rescue medication use). The theoretical range of AUC0-72 is 0-720.
Time Frame: 72 hours
Population: ITT Population
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Cohort 1, Group 1: HTX-011 | Cohort 1, Group 2: HTX-011 | Cohort 1, Group 3: Saline Placebo | Cohort 1, Group 4: Bupivacaine HCI | Cohort 2, Group 1: HTX-011 | Cohort 2, Group 2: HTX-011 + Ropivacaine | Cohort 2, Group 3: Saline Placebo | Cohort 2, Group 4: Bupivacaine HCI
Number analyzed (Participants) | 20 | 22 | 11 | 10 | 58 | 56 | 53 | 55
pain intensity score*hr | 543.14 (142.566) | 560.85 (136.099) | 576.44 (150.815) | 468.58 (179.687) | 471.19 (149.443) | 452.54 (194.095) | 577.93 (125.102) | 516.93 (152.512)

3. Secondary Outcome: Mean Total Postoperative Opioid Consumption (in Morphine Equivalents)
Time Frame: 72 hours
Population: ITT Population
Measure: Mean (Standard Deviation); unit: morphine milligram equivalent (MME)
Groups:
- Cohort 2, Group 1: HTX-011: HTX-011, 400 mg/12 mg via instillation.
- Cohort 2, Group 2: HTX-011 + Ropivacaine: HTX-011, 400 mg/12 mg via instillation; Ropivacaine, 50 mg via injection.
Arm/Group | Cohort 1, Group 1: HTX-011 | Cohort 1, Group 2: HTX-011 | Cohort 1, Group 3: Saline Placebo | Cohort 1, Group 4: Bupivacaine HCI | Cohort 2, Group 1: HTX-011 | Cohort 2, Group 2: HTX-011 + Ropivacaine | Cohort 2, Group 3: Saline Placebo | Cohort 2, Group 4: Bupivacaine HCI
Number analyzed (Participants) | 20 | 22 | 11 | 10 | 58 | 56 | 53 | 55
morphine milligram equivalent (MME) | 65.53 (31.615) | 66.86 (31.154) | 70.41 (18.057) | 60.70 (29.903) | 64.39 (27.889) | 60.32 (34.949) | 73.55 (34.448) | 68.35 (29.169)

ADVERSE EVENTS:
Time Frame: 28 Days.
Description: Subjects reporting more than one TEAE are counted only once.
Groups:
- Cohort 1, Group 2: HTX-011: HTX-011 (bupivacaine/meloxicam), 200 mg/6 mg via injection and instillation(combination).
Arm/Group | Cohort 1, Group 1: HTX-011 | Cohort 1, Group 2: HTX-011 | Cohort 1, Group 3: Saline Placebo | Cohort 1, Group 4: Bupivacaine HCI | Cohort 2, Group 1: HTX-011 | Cohort 2, Group 2: HTX-011 + Ropivacaine | Cohort 2, Group 3: Saline Placebo | Cohort 2, Group 4: Bupivacaine HCI
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22 | 0/11 | 0/10 | 0/58 | 0/56 | 0/53 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/22 | 0/11 | 1/10 | 1/58 | 4/56 | 3/53 | 2/55
Other Adverse Events (participants affected / at risk) | 19/20 | 22/22 | 11/11 | 10/10 | 55/58 | 50/56 | 50/53 | 49/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Group 1: HTX-011 (N=20) | Cohort 1, Group 2: HTX-011 (N=22) | Cohort 1, Group 3: Saline Placebo (N=11) | Cohort 1, Group 4: Bupivacaine HCI (N=10) | Cohort 2, Group 1: HTX-011 (N=58) | Cohort 2, Group 2: HTX-011 + Ropivacaine (N=56) | Cohort 2, Group 3: Saline Placebo (N=53) | Cohort 2, Group 4: Bupivacaine HCI (N=55)
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Group 1: HTX-011 (N=20) | Cohort 1, Group 2: HTX-011 (N=22) | Cohort 1, Group 3: Saline Placebo (N=11) | Cohort 1, Group 4: Bupivacaine HCI (N=10) | Cohort 2, Group 1: HTX-011 (N=58) | Cohort 2, Group 2: HTX-011 + Ropivacaine (N=56) | Cohort 2, Group 3: Saline Placebo (N=53) | Cohort 2, Group 4: Bupivacaine HCI (N=55)
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 5 | 2 | 1 | 4 | 6 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 1 | 3 | 6 | 4 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 2 | 1 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 0 | 0 | 1 | 6 | 6 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 4 | 4 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 5 | 5 | 4 | 3 | 9 | 8 | 9 | 8
Headache (Nervous system disorders) | 3 | 3 | 2 | 1 | 4 | 2 | 0 | 4
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 4 | 4 | 1 | 0 | 9 | 9 | 11 | 6
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 3 | 1 | 4 | 11 | 8 | 8 | 7
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 3 | 2 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 | 16 | 6 | 4 | 29 | 30 | 25 | 30
Constipation (Gastrointestinal disorders) | 8 | 10 | 2 | 3 | 14 | 21 | 12 | 18
Vomiting (Gastrointestinal disorders) | 7 | 6 | 4 | 2 | 15 | 14 | 10 | 15
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 2 | 3 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 4 | 4 | 1 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 2 | 5 | 2 | 5 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 2 | 1 | 0 | 3 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 4 | 4 | 6 | 2
Pyrexia (General disorders) | 1 | 5 | 0 | 2 | 8 | 8 | 2 | 8
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 0
Medical device site reaction (General disorders) | 0 | 0 | 0 | 2 | 3 | 2 | 1 | 1
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Oedema peripheral (General disorders) | 2 | 3 | 0 | 1 | 1 | 0 | 3 | 1
Peripheral swelling (General disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 4 | 3 | 2 | 1 | 0 | 2 | 5 | 1
Wound drainage (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incision site oedema (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1 | 7 | 3 | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT03015532/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT03015532/SAP_001.pdf